CLINICAL TRIAL: NCT04706364
Title: Investigations of Sensorimotor Plasticity in Autism Spectrum Disorders
Brief Title: Investigation of Brain Plasticity in Autism Spectrum Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Simons Foundation Autism Research Initiative (SFARI) (Unknown)
Responsible Party: Principal Investigator, Alexander Rotenberg, Associate Professor of Neurology, Boston Children's Hospital
Other Study IDs: IRB-P00027556; R21MH120438 (NIH)
Record Dates: First submitted 2021-01-11; First posted 2021-01-12 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Neuropsychological Tests; Electroencephalography; Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva sample for genetic testing (optional)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder (ASD): Individuals diagnosed with an Autism Spectrum Disorder
  Interventions: Behavioral: Neuropsychological Testing; Genetic: (Optional) Saliva Collection; Device: Sensory Testing; Device: Electroencephalogram (EEG); Device: Transcranial Magnetic Stimulation
- Healthy Control: Typically developing individuals without a history of autism
  Interventions: Behavioral: Neuropsychological Testing; Genetic: (Optional) Saliva Collection; Device: Sensory Testing; Device: Electroencephalogram (EEG); Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Behavioral: Neuropsychological Testing — Includes an IQ test, Autism Diagnostic Observation Schedule-2 (ADOS-2), and Autism Diagnostic Interview-Revised (ADI-R) assessments.
Genetic: (Optional) Saliva Collection — The sample is to test for genes (BDNF/APOE/COMT) that everyone has, but people have different varieties of these genes.
  Genetic testing is funded by Boston Children's Hospital.
Device: Sensory Testing — Three different tests will be completed:
  the tactile prepulse inhibition test (PPI) texture perception indentation testing (Mechanical Detection Threshold).
  Investigators will also apply mild electrical stimulation to the median nerve of the hand (on the wrist).
  The second sensory visit will be another version of the PPI testing involving hearing and sound.
Device: Electroencephalogram (EEG) — A cap will be placed on the participants head that will be filled with electrodes (small discs). The EEG will allow investigators to measure how the brain reacts to the sensory testing.
Device: Transcranial Magnetic Stimulation — Single pulses of TMS, as well as PAS (a second type of TMS), will be applied to the cortex.
  There will be two - four identical TMS testing visits.

SUMMARY:
Individuals with autism spectrum disorders (ASD) commonly experience variances in tactile behaviors, such as hypersensitivity to light touch stimuli, altered texture discrimination, and hyporesponsivity to pain. Researchers aim to investigate the somatosensory sensitivity and sensorimotor integration utilizing novel, objective behavioral assays and TMS. The main purpose is to study brain plasticity (the changes that occur in the brain through experience) in individuals with autism spectrum disorders.

DETAILED DESCRIPTION:
Individuals with autism spectrum disorders (ASD) commonly experience variances in tactile behaviors, such as hypersensitivity to light touch stimuli, altered texture discrimination and hyporesponsivity to pain. The degree of this somatosensory impairment correlates with increased anxiety behaviors as well as impairments in social behavior among ASD patients.

There remains an unmet need for suppressing the tactile hypersensitivity, which may improve anxiety and other core symptoms of ASD; however, methodologies for measuring tactile sensitivity vary widely across clinical and basic research fields. There is an urgent need for direct and objective sensory reactivity metrics in clinical studies to assess deficits in specific patient populations and for designing effective therapeutic strategies. As compared with traditional behavioral methods, the investigators propose to test novel, objective and quantitative metrics of somatosensory sensitivity in individuals with ASD.

In addition, transcranial magnetic stimulation (TMS) provides a method of measuring cortical reactivity offering the advantage of providing behaviorally independent results that are largely unaffected by attention or cognitive ability. Therefore, a TMS-based physiologic biomarker may be applicable to all individuals across the autism spectrum. A form of TMS known as paired associative stimulation (PAS) can be used to study the suggested impairment in integration of sensory input into cortical function that underlies tactile hypersensitivity in ASD. Thus, the investigators aim to investigate somatosensory sensitivity and sensorimotor integration utilizing novel, objective behavioral assays and TMS.

Participation in the study will consist of up to seven visits: one screening visit, two sensory testing visits, and two - four TMS sessions. The screening visit is expected to last between 2-3 hours, during which participants will first provide informed consent. Participants will then receive a thorough medical examination by a neurologist, and a neuropsychological evaluation (including IQ measures and ASD specific evaluations). If eligible to continue, participants will then come back for two sensory visits and two - four TMS visits that are spaced a minimum of 1 week apart.

ELIGIBILITY:
Inclusion Criteria:

* For ASD group:

  * Clinical diagnosis of a disorder on the autism spectrum according to:

    1. DSM-IV or DSM 5 criteria
    2. IQ>70 (as determined by the Abbreviated Stanford-Binet IQ)
* For the Control group:

  * No history of ASD or other developmental delay
  * No history of ASD or other developmental delay in first-degree relatives.
  * No history of clinical diagnosis of an anxiety disorder

Exclusion Criteria:

* Both ASD and Control groups:

  * Intracranial pathology, cerebral palsy, history of severe head injury, or syndromic dysmorphology
  * History of fainting spells of unknown or undetermined etiology that might constitute seizure
  * History of seizure or epilepsy
  * Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency
  * Metal implants (excluding dental fillings) or devices such as pacemaker, medication pump, nerve stimulator, TENS unit, ventriculo-peritoneal shunt unless cleared by the responsible MD
  * Substance abuse or dependence within the past six months
  * Chronic treatment with prescription medications that decrease cortical seizure threshold
  * Peripheral neuropathy, as determined by the study MD during neurologic exam
* For the Control group:

  * For control participants' medical history will be reviewed for diagnoses of neurologic or psychiatric disease. If in the judgment of the investigator, the condition, e.g., depression, is well-controlled with stable medications, and does not include abnormalities of the sensory motor systems, they may be included in the study. Control participants will be excluded from taking part in the study if they have a 1st degree relative with ASD.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children diagnosed with an Autism Spectrum Disorder (ASD), as well as controls.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Textured novel object recognition test (NORT) and mechanical detection threshold (MDT) with von Frey hairs | 3 years
  To assess the validity of tactile prepulse inhibition (PPI) and other quantitative somatosensory assessments as potential biomarkers for somatosensory dysfunction in children with ASD. These metrics will provide a valuable comparison to the more-quantitative physiological measures by PAS and PPI.
Somatosensory temporal discrimination threshold (STDT) and PAS-induced modulation of motor-evoked potentials (MEPs) | 3 years
  To assess the validity of PAS-induced modulation of corticospinal excitability as a neurophysiologic biomarker for somatosensory dysfunction in children with ASD.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rotenberg, MD, PhD, Principal Investigator — Alexander.Rotenberg@childrens.harvard.edu
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States